CLINICAL TRIAL: NCT05521100
Title: Comparison of Safety and Efficacy Between the Application of Vascular Closure Device and Conventional Figure-of-eight Suture in Transvenous Cardiac Interventional Surgery
Brief Title: Application of Vascular Closure Device in Transvenous Cardiac Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Director of Cardiology, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSH-ACT
Record Dates: First submitted 2022-08-29; First posted 2022-08-30 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Vascular Access Complications
MeSH Terms: interventions — Vascular Closure Devices

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proglide group (Experimental): Vascular Sutures for Transvenous Cardiac Interventions Using Proglide
  Interventions: Procedure: Vascular closure device
- figure eight stitch (Active Comparator): Vascular Sutures for Transvenous Cardiac Intervention Using Conventional Figure-8 Sutures
  Interventions: Procedure: figure eight stitch

INTERVENTIONS:
Procedure: Vascular closure device — Suture of lower extremity veins using the Proglide Vascular Closure Device
  Arms: Proglide group
Procedure: figure eight stitch — Vascular Sutures for Transvenous Cardiac Intervention Using Conventional Figure-8 Sutures
  Arms: figure eight stitch

SUMMARY:
Comparison of safety and efficacy between the application of vascular closure device and conventional figure-of-eight suture in transvenous cardiac interventional surgery

DETAILED DESCRIPTION:
Comparison of safety and efficacy between the application of vascular closure device and conventional figure-of-eight suture in transvenous cardiac interventional surgery.From the operation success rate, postoperative bleeding, immobilization time, the rate of revisiting the doctor due to wound problems within 1 month, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving lower extremity venous intervention with a diameter of 12F or more

Exclusion Criteria:

* None

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Vascular bleeding event rate | 1month
  Proportion of bleeding after two methods of vascular suturing

SECONDARY OUTCOMES:
bed braking time | 1 day
  Postoperative bed rest time

CONTACTS AND LOCATIONS:
Overall Officials: Yawei Xu, PhD, Study Chair — Tongji University
Locations (1):
- Jun Zhang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No